CLINICAL TRIAL: NCT03885180
Title: Randomized Evaluation of D-dimer Guiding Duration of Oral Anticoagulation Therapy in Patients With Bioprosthetic Heart Valves
Brief Title: Randomized Evaluation of D-dimer Guiding dUration of Oral antiCoagulation thErapy
Acronym: REDUCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Principal Investigator, Litao Zhang, MD, Head of anticoagulation clinic, Wuhan Asia Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-P-026
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Valve Heart Disease; Anticoagulants; Increased
Keywords: bioprosthetic heart valves; oral anticoagulation; thrombotic events
MeSH Terms: conditions — Heart Valve Diseases | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extend anticoagulation group (Experimental): Extended the duration anticoauglation to 12 months
  Interventions: Drug: Warfarin Sodium
- Stop anticoagulation group (No Intervention): Just stop oral anticoagulation like routine

INTERVENTIONS:
Drug: Warfarin Sodium — Extending warfarin anticoagulation
  Arms: Extend anticoagulation group

SUMMARY:
Guidelines recommended that patients with bioprosthetic heart valves (BHV) only need 6 months oral anticoagulation therapy after operation. However, a small part of patients still suffered thrombotic events after withdrawal of warfarin, which means these patients may need extend anticoagulation therapy. D-dimer, a sensitive marker of thrombosis or prethromboembolism state. Previous studies have demostrated that patients with elevated D-dimer levels have significant more clinical outcomes than those with nagative D-dimer levels. The aim of this study was to evaluate whether D-dimer could guide the duration of oral anticoagulation therapy in patients with BHV.

DETAILED DESCRIPTION:
Patients with BHV were screened and enrolled in this study. D-dimer levels were measured in the sixth months after BHV operation but before withdrawal of warfarin. Patients with elevated D-dimer were randomized to extend anticoagulation therapy group and routine stopping anticoagulation group.

ELIGIBILITY:
Inclusion Criteria:

* Patients received BHV within 3 months

Exclusion Criteria:

* Recently throboemblism within 6 months
* Recently bleedings within 3 months
* Evaluated lifetime less than 2 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Thrombotic events | 24 months
  Stroke, DVT, PE, valve thrombosis
Bleeding events | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Asia Heart Hospital, Wuhan, Hubei, China